CLINICAL TRIAL: NCT01170806
Title: Study of Pharmacodynamic Equivalence of Two Commercial Formulations of Orlistat (Lipiblock vs Xenical) on Intestinal Lipases Inhibition
Brief Title: Study of Fat Malabsorption by Lipiblock Versus Xenical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Germed Pharma (Industry)
Responsible Party: Bruno Geloneze, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LIMED0008
Record Dates: First submitted 2010-05-18; First posted 2010-07-27 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: Intestinal lipase; Orlistat; fecal fat; obesity
MeSH Terms: conditions — Obesity | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orlistat (Lipiblock) treatment (Active Comparator): Lipiblock is a new Orlistat formulation, produce by Germed Pharma, Brazil. Capsule 120mg
  Interventions: Drug: Orlistat
- Orlistat (Xenical) treatment (Active Comparator): Xenical is a innovator Orlistat formulation, produced by Roche
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — Capsules of 120mg of two commercial formulations of Orlistat (Lipiblock or Xenical) were taken 3 times daily for 7 dayy
  Other Names: Xenical; Lipiblock; Tetrahydrolipstatin

SUMMARY:
Obesity is a chronic condition with fat-rich diets playing a major role in its etiology. Pharmacological therapy has been proposed for weight loss and maintenance. This study aims to study the intestinal lipase blockade by partial inhibition of fat absorption after treatment with two commercials formulations of Orlistat.

DETAILED DESCRIPTION:
The overweight and obesity epidemic affects approximately 1.6 millions of people worldwide. Obesity is a chronic condition, associated with premature death, co-morbidities, risk factors for main cardiac disease, stigmatization and significant economic costs. The causes of obesity are complex and include the interplay of environmental, social, economic and genetic factors. Besides fat-rich diets also play a significant role in the etiology of obesity. Correct diet orientation associated with physical exercise usually did not lead to expected result in weight loss and maintenance. Pharmacological therapy has been proposed as an adjunct to achieve the ideal weight. Orlistat acts in reduction of lipids absorption by inhibition of gastric and pancreatic lipases in gastrointestinal tract leading to sustained weight loss. This is a double blind study, randomized, of 2 weeks. The aim of this study was evaluate the intestinal lipase blockade by decrease of fat absorption of fecal fat after treatment with two commercials formulations of Orlistat in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* BMC (Body Mass Index) between 30 to 40 kg/m2
* Women
* 18 to 45 years
* Premenopausal stage

Exclusion Criteria:

* Relevant diseases (diabetes, cardiovascular, gastrointestinal, renal and hepatic diseases, endocrine disorders, hemoglobinopatHy or neoplasm in the last three years)
* Chemical or natural laxatives
* Weight variation greater than 5% in the preceding 3 months
* Surgery for weight reduction
* Drugs to obesity control and/or oral corticosteroids anti-inflammatory in the last three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Study of equivalence between two commercial capsules of Orlistat on fat absorption inhibition | baseline
  This study aim to investigate differences in fat absorption inhibition after 7 days treatment with Lipiblock and Xenical (two commercial capsules of Orlistat). Therefore, total fecal fat and fecal fat percentage wil be analysed, comparing these data before and after treatment with Lipiblock and Xeical.

SECONDARY OUTCOMES:
Study of equivalence between two commercial capsules of Orlistat on fat absorption inhibition | after 7 days Orlistat treatment
  This study aim to investigate differences in fat absorption inhibition after 7 days treatment with Lipiblock and Xenical (two commercial capsules of Orlistat). Therefore, total fecal fat and fecal fat percentage wil be analysed, comparing these data before and after treatment with Lipiblock and Xenical.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, MD PhD, Principal Investigator — University of Campinas (UNICAMP); Sabrina Nagassaki, PharmD PhD, Study Chair — University of Campinas (UNICAMP); Christiane Stabe, MSc, Study Chair — University of Campinas (UNICAMP); Daniela Tezoto, Study Chair — University of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/University of Campinas (UNICAMP), Campinas, São Paulo, Brazil